CLINICAL TRIAL: NCT05105308
Title: Chompions! A Treatment Study for Childhood Avoidant/Restrictive Food Intake Disorder (ARFID)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00103645; 1R33MH121549-01A1 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: ARFID; Picky Eating; Eating Disorders in Children
Keywords: FBI-ARFID; Eating Disorder; Avoidant Restrictive Food Intake Disorder; Food Neophobia; Treatment for Children; Sensory Sensitivity; Picky Eating; Low Weight; Nutritional Deficiencies
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Food Fussiness; Feeding and Eating Disorders; Thinness; Malnutrition | interventions — Flavin-Adenine Dinucleotide

STUDY DESIGN:
Intervention Model Description: The design is a two-group (n=70 per group) randomized controlled trial. Primary outcomes including ARFID symptoms and secondary outcomes (e.g., responder status of weight gain) will be assessed at baseline, posttreatment, and 3-month follow-up, while abbreviated measures will be assessed every session.
Who Masked: Outcomes Assessor
Masking Description: Individuals who conduct the diagnostic interview will not be informed of the intervention arm to which a child is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Assisted Diet (FAD) (Active Comparator): This is a 20-session intervention with a child and the child's parents that consists of helping parents set goals around their child's renourishment; consider barriers to implementing proposed plans; thinking through strategies to avoid barriers; and providing ongoing support for plan implementation.
  Interventions: Behavioral: Family Assisted Diet (FAD)
- Feeling and Body Investigator_ARFID Division (FBI-ARFID) (Experimental): This is a 20-session intervention with a child and the child's parents that consists of 4 components: 1) psychoeducation of somatic body sensations and sensory features of foods using playful characters (e.g., Aftertaste Anthony); 2) in-session exercises that expose family members to different body and food sensations so they can learn something new about their body and food; 3) body brainstorm worksheets that help them generalize what they learn in session to outside of treatment; and 4) Decision-tree practice worksheets that help them map body sensations to meanings and actions and to track explorations with food.
  Interventions: Behavioral: Feeling and Body Investigator_ARFID Division (FBI-ARFID)

INTERVENTIONS:
Behavioral: Family Assisted Diet (FAD) — A behavioral intervention consisting of helping parents renourish their child and conduct food exposures with new foods.
  Other Names: FAD
  Arms: Family Assisted Diet (FAD)
Behavioral: Feeling and Body Investigator_ARFID Division (FBI-ARFID) — A sensory and somatic focused intervention that educates children about feelings and bodily sensations, in-session exposures to body and food sensations, different strategies to improve generalization while at home, and strategies to help them understand and track experiences exploring food.
  Other Names: FBI-ARFID
  Arms: Feeling and Body Investigator_ARFID Division (FBI-ARFID)

SUMMARY:
Avoidant Restrictive Food Intake Disorder (ARFID) is a disorder that affects toddlers, children, adolescents, and adults. Individuals with ARFID are not able to consume an adequate amount or variety of food to a degree that it affects their mental and/or physical health. ARFID often begins in early childhood so it is important to treat children in early in life as possible to prevent any negative consequences of poor nutrition. There are currently no treatments for young children with ARFID. The investigators have developed two different study programs and the purpose of this study is to test them out and see if they help children with ARFID and to learn more about how these study programs work.

ELIGIBILITY:
Inclusion Criteria:

* Child is between 60 and 119 months (5 years and up to 9 years, 11 months)
* English Speaking
* Consent given by parent and assent by child

And any one or more of the following:

* Score of 29 or above on the Child Food Neophobia Scale
* Underweight
* Current diagnosis of ARFID
* Dependent on nutritional supplements to achieve sufficient calories for optimal growth
* Avoiding activities due to eating rated at least almost always

Exclusion Criteria:

* Child is known to have a severe intellectual disability based on medical chart review
* Meets diagnostic criteria for anorexia nervosa or bulimia nervosa
* Is currently enrolled in a treatment study or receiving active treatment for ARFID
* Taking medications known to affect appetite

Ages: 60 Months to 119 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-11-19 (Estimated)

PRIMARY OUTCOMES:
Change in the number of clinically severe symptoms of Avoidant Restrictive Food Intake Disorder (ARFID) as measured by the PARDI (Pica, ARFID, and Rumination Diagnostic Interview) | Baseline, Post-Treatment (up to 30 weeks), 3-Months Post-Treatment
  The 17-item PARDI measures symptoms including body mass index, diet quality, dependence on supplement use for sufficient calories, and psychosocial impairment. Each item assesses a symptom on a 0 - 6 scale, with scores above 4 indicating that it is a clinically severe symptom.

SECONDARY OUTCOMES:
Nutrition Quantity as measured by 3-day 24-hour dietary recalls | Baseline
  Nutrition Quantity is measured by two weekdays and one weekend day assisted dietary recall with the parent of the child. Using the Harris-Benedict equation to determine a child's nutritional needs, the following will be measured: 1) Child unable to meet daily energy requirements without supplement and/or 2) Child's dietary intake is below energy needs on all 3 days.
Nutrition Quantity as measured by 3-day 24-hour dietary recalls | Post-Treatment (up to 30 weeks)
  Nutrition Quantity is measured by two weekdays and one weekend day assisted dietary recall with the parent of the child. Using the Harris-Benedict equation to determine a child's nutritional needs, the following outcomes will be measured: 1) Child unable to meet daily energy requirements without supplement and/or 2) Child's dietary intake is below energy needs on all 3 days.
Psychosocial Functioning as measured by items on the PARDI | Baseline
  Psychosocial functioning is measured by items on the PARDI indicating that the child does not avoid social events due to eating/food and less than or equal to 1 indicating that the child is able to remain at the table and demonstrate age-appropriate behaviors.
Psychosocial Functioning as measured by items on the PARDI | Post-Treatment (up to 30 weeks)
  Psychosocial functioning is measured by items on the PARDI indicating that the child does not avoid social events due to eating/food and less than or equal to 1 indicating that the child is able to remain at the table and demonstrate age-appropriate behaviors.
Psychosocial Functioning as measured by items on the PARDI | 3-Months Post-Treatment
  Psychosocial functioning is measured by items on the PARDI indicating that the child does not avoid social events due to eating/food and less than or equal to 1 indicating that the child is able to remain at the table and demonstrate age-appropriate behaviors.
Nutrition Quality as measured by 3-day 24-hour dietary recalls | Baseline
  Nutrition Quality is measured by the average macronutrient and micronutrient assessment from two weekdays and one weekend day assisted dietary recall with the parent of the child.
Nutrition Quality as measured by 3-day 24-hour dietary recalls | Post-Treatment (up to 30 weeks)
  Nutrition Quality is measured by the average macronutrient and micronutrient assessment from two weekdays and one weekend day assisted dietary recall with the parent of the child.
Body Mass Index (BMI) as measured by height and weight | Baseline
  BMI will be measured by parents at home with scales and tape measures provided to them.
Body Mass Index (BMI) as measured by height and weight | Weekly (up to 30 weeks)
  BMI will be measured by parents at home with scales and tape measures provided to them.
Body Mass Index (BMI) as measured by height and weight | Post-Treatment (up to 30 weeks)
  BMI will be measured by parents at home with scales and tape measures provided to them.
Body Mass Index (BMI) as measured by height and weight | 3-Months Post-Treatment
  BMI will be measured by parents at home with scales and tape measures provided to them.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Zucker, PhD, Principal Investigator — Duke University; Guillermo Sapiro, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucker N, Mauro C, Craske M, Wagner HR, Datta N, Hopkins H, Caldwell K, Kiridly A, Marsan S, Maslow G, Mayer E, Egger H. Acceptance-based interoceptive exposure for young children with functional abdominal pain. Behav Res Ther. 2017 Oct;97:200-212. doi: 10.1016/j.brat.2017.07.009. Epub 2017 Jul 29. PMID 28826066
- [Background] Zucker NL, LaVia MC, Craske MG, Foukal M, Harris AA, Datta N, Savereide E, Maslow GR. Feeling and body investigators (FBI): ARFID division-An acceptance-based interoceptive exposure treatment for children with ARFID. Int J Eat Disord. 2019 Apr;52(4):466-472. doi: 10.1002/eat.22996. Epub 2018 Dec 31. PMID 30597590

DOCUMENTS (1):
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT05105308/ICF_000.pdf